CLINICAL TRIAL: NCT03724422
Title: Prophylaxis Low-Dose Radiation Therapy for Heterotopic Ossification in Distal Humerus Fractures
Brief Title: HO Prophylaxis Therapy for Distal Humerus Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty getting radiation therapy for patients and Low enrollment number
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Rodolfo Zamora, MD, Assistant Professor of Orthopaedic Surgery, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB Number:18.0184
Record Dates: First submitted 2018-09-20; First posted 2018-10-30 (Actual); Results first posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Heterotopic Ossification; Humeral Fractures; Radiation Therapy
Keywords: Herteropic Ossification
MeSH Terms: conditions — Ossification, Heterotopic; Humeral Fractures | interventions — Radiation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either a treatment or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): This group will receive the standard of care treatment for their distal humerus fracture only.
- Intervention (Experimental): This group will receive the prophylactic radiation therapy in addition to the standard of care treatment of their distal humerus fracture.
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — A dose of 500cGy will be delivered in 1 fraction to the isocenter. Radiation will be administered no later than 72 hours postoperatively
  Arms: Intervention

SUMMARY:
To determine the effectiveness of 500 cGy dose of radiation therapy vs. an untreated group in the prophylactic treatment of heterotopic ossification in distal humerus fractures

DETAILED DESCRIPTION:
Heterotopic ossification is the formation of ectopic lamellar bone in the soft tissues. The process is thought to occur through local and distal recruitment osteoprogenitor cells especially mesenchymal stem cells which lead to HO formation based on local microenvironmental factors including activation of the BMP-mediated pathways.1 There are several risk factors associated with HO development such as central nervous system injury, thermal burn, hip arthroplasty, acetabular fractures, and elbow fractures; HO is also seen with certain arteriopathies and genetic conditions e.g. ankylosing spondylitis, seronegative arteriopathies, diffuse idiopathic skeletal hyperostosis (DISH), and fibrodysplasia ossificans progressive. In elbow fractures, the prevalence of HO is around 40%, and of those that develop HO, 20% experience a clinically relevant decrease in elbow range of motion with a flexion-extension arc of <100°. In a study by Foruria, et al. of 89 patients with a distal humerus fracture without associated proximal radius or ulna fracture that underwent surgical treatment with ORIF, 42% developed HO and the HO in these patients was associated with significantly less extension and a limited flexion-extension arc but was not associated with a change in supination or pronation. Abrams, et al. looked at the development of HO after elbow fracture fixation in 89 pts including 20 distal humerus fractures and found that distal humeral fractures were more likely to have higher grade of HO, have more compromised functional outcomes, and require return to the OR more often for capsular release with HO resection at a rate of 25%. Prophylactic treatment for HO is most commonly achieved through the use of NSAIDs such as indomethacin and radiation therapy. Both modalities have the risk of nonunion of fracture and radiation therapy has additional risks such as delayed wound healing, soft tissue contracture, and the theoretical risk of malignancy although no cases of malignancy after prophylactic radiation have been reported to date. Radiation therapy in the prevention of HO has been well studied in the hip with low-dose radiation being established as an effective dose and 700cGy as the most commonly used dose.5 Radiation therapy in the prevention of HO at the elbow is not as well studied and existing studies have commonly used a dose of 700cGy. One study looked at the use of radiation therapy in combination of patients being treated acutely for elbow trauma and patients being treated for HO after previous elbow trauma, and the study found that 3 of the 36 patients developed new HO and found an occurrence of 2 nonunion with the majority treated with 700cGy but 2 pts received 600cGy.6 Heyd, et al. present a case series of 9 patients that underwent surgical excision of clinically significant HO at the elbow and received radiation therapy of 2 doses of 500cGy, 1 dose of 600 cGy , or 1 dose of 700 cGy ; at a mean follow up of 7.7 no patients had recurrence of HO and 8 of 9 showed clinical improvement.7 A study of 11 patients that underwent ORIF for fracture-dislocation of the elbow and single-dose radiation therapy of 700 cGy within 72 hours postoperatively, and 3 patients (27%) developed radiographic evidence of HO while 10 patients (91%) had no functional limitations and 100% of patients completely healed there fracture without complications at average follow up of 12 months (9-24 months). 3 of the 11 patients had distal humerus fractures and none of them had radiographic evidence of HO or functional limitation.8 A recent multicenter randomized control trial of patients with intraarticular distal humerus fractures or fracture-dislocation of the elbow with proximal ulna and/or radius fracture randomized patients to either receive a single dose of 700cGy within 72 hours postop or receive nothing for HO prophylaxis. Although, HO occurrence in the 21 patients in the treatment group vs the 24 in the control group (33% vs 54%), the rate of nonunion was higher in the treatment group (38% vs 4%) resulting in termination of the study. Several studies have demonstrated the efficacy and safety of radiation therapy in the prophylactic treatment of HO in the elbow, but the study by Hamid questions the use of a 700 cGy dose because of the rate of nonunion observed. Thus, the investigators hypothesize that a dose of 500 cGy will be adequate in the elbow HO prevention as there is smaller treatment area compared to the hip where 700 cGy is an effective dose and that this dose will not result in an increased rate of nonunion.

Early osteoprogenitor cells involved in bone repair are thought to be more radiosensitive than the more mature cells seen later in the development of bone formation after fracture. Thus, radiation specifically works to inhibit the osteogenic pathway. Based on a recent Cochrane review, the incidence of HO development with any dose of RT was 24%. The was no correlation with site (hip, elbow, knee) or radiation dose, which ranged from 500cGy - 2000cGy. The most commonly used regimen was 700cGy (60%) while dose less than 700cGy represented 12%. The problem with 700cGy is the reported rate of non-union is as high as 40%, especially when the elbow is treated. Additionally, increasing radiation dose alters the expression of transforming growth factor-beta 1, vascular endothelial growth factor, and alkaline phosphatase which can prevent bone union. Based on this data, 500cGy should still be adequate to inhibit the osteogenic pathway by causing lethal damage to osteoprogenitor cells while at the same potentially allowing for a better bone union.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a distal humerus fracture.
2. Patient's age is greater than or equal to 18

Exclusion Criteria:

1. Patient has a concomitant proximal ulna and/or proximal radius fracture
2. Patient requires external fixation of the elbow
3. Patient has quadriplegia or paraplegia
4. Patient requires intubation upon admission or for >4 hours during admission for nonsurgical purposes
5. Patient has concomitant soft tissue damage in the affected elbow that cannot be appropriately closed within 72 hours of surgery
6. Patient has a burn affecting greater than or equal to 20% of the total body surface area or on the affected elbow
7. Patient has pre-existing heterotopic ossification in the affected elbow.
8. Patient is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Zamora, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
No plan at this time to Share IPD

REFERENCES:
- [Background] Ranganathan K, Loder S, Agarwal S, Wong VW, Forsberg J, Davis TA, Wang S, James AW, Levi B. Heterotopic Ossification: Basic-Science Principles and Clinical Correlates. J Bone Joint Surg Am. 2015 Jul 1;97(13):1101-11. doi: 10.2106/JBJS.N.01056. PMID 26135077
- [Background] Kaplan FS, Glaser DL, Hebela N, Shore EM. Heterotopic ossification. J Am Acad Orthop Surg. 2004 Mar-Apr;12(2):116-25. doi: 10.5435/00124635-200403000-00007. PMID 15089085
- [Background] Foruria AM, Lawrence TM, Augustin S, Morrey BF, Sanchez-Sotelo J. Heterotopic ossification after surgery for distal humeral fractures. Bone Joint J. 2014 Dec;96-B(12):1681-7. doi: 10.1302/0301-620X.96B12.34091. PMID 25452373
- [Background] Abrams GD, Bellino MJ, Cheung EV. Risk factors for development of heterotopic ossification of the elbow after fracture fixation. J Shoulder Elbow Surg. 2012 Nov;21(11):1550-4. doi: 10.1016/j.jse.2012.05.040. Epub 2012 Sep 2. PMID 22947234
- [Background] Davis JA, Roper B, Munz JW, Achor TS, Galpin M, Choo AM, Gary JL. Does Postoperative Radiation Decrease Heterotopic Ossification After the Kocher-Langenbeck Approach for Acetabular Fracture? Clin Orthop Relat Res. 2016 Jun;474(6):1430-5. doi: 10.1007/s11999-015-4609-y. PMID 26497882
- [Background] Robinson CG, Polster JM, Reddy CA, Lyons JA, Evans PJ, Lawton JN, Graham TJ, Suh JH. Postoperative single-fraction radiation for prevention of heterotopic ossification of the elbow. Int J Radiat Oncol Biol Phys. 2010 Aug 1;77(5):1493-9. doi: 10.1016/j.ijrobp.2009.06.072. PMID 20637977
- [Background] Heyd R, Strassmann G, Schopohl B, Zamboglou N. Radiation therapy for the prevention of heterotopic ossification at the elbow. J Bone Joint Surg Br. 2001 Apr;83(3):332-4. doi: 10.1302/0301-620x.83b3.11428. PMID 11341414
- [Background] Stein DA, Patel R, Egol KA, Kaplan FT, Tejwani NC, Koval KJ. Prevention of heterotopic ossification at the elbow following trauma using radiation therapy. Bull Hosp Jt Dis. 2003;61(3-4):151-4. PMID 15156818
- [Background] Hamid N, Ashraf N, Bosse MJ, Connor PM, Kellam JF, Sims SH, Stull DE, Jeray KJ, Hymes RA, Lowe TJ. Radiation therapy for heterotopic ossification prophylaxis acutely after elbow trauma: a prospective randomized study. J Bone Joint Surg Am. 2010 Sep 1;92(11):2032-8. doi: 10.2106/JBJS.I.01435. PMID 20810853

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention
Started | 1 | 2
Completed | 1 | 0 (Patients had interval healing then lost follow up)
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 | 42 (25.46) | 44.3 (18.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 32.7 | 30.6 (16.97) | 31.3 (12.06)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Presence of HO on Humerus
Description: Presence of heterotopic ossification on plain radiographs taken in the anteroposterior and lateral planes within 1 year after surgery as quantified using the classification systems described by Brooker, et al. and Hastings and Graham
Time Frame: 1 year. The control patient completed 366 days of follow up. The two intervention patients lost follow up after 155 days and 62 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

2. Secondary Outcome: Non-union at the Fracture Site.
Description: Rate of non-union of both groups requiring revision surgery.
Time Frame: 1 year post surgical reduction. The control patient completed 366 days of follow up. The two intervention patients lost follow up after 155 days and 62 days respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT03724422/Prot_001.pdf